CLINICAL TRIAL: NCT00093301
Title: Efficacy of Levosimendan in the Critically Ill Patients With Unstable Hemodynamics (the LICI Study) - A Double Blind Randomized Pilot Study
Brief Title: Levosimendan Versus Dobutamine in Shock Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wentworth Area Health Services (Other)
Collaborators: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03/007
Record Dates: First submitted 2004-10-05; First posted 2004-10-07 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-10

CONDITIONS: Cardiogenic Shock; Septic Shock
Keywords: Shock; Levosimendan; Inotropes; Dobutamine; Heart failure; Sepsis
MeSH Terms: conditions — Shock, Cardiogenic; Shock, Septic; Shock; Heart Failure; Sepsis | interventions — Simendan; Dobutamine

INTERVENTIONS:
Drug: Levosimendan
Drug: Dobutamine

SUMMARY:
The purpose of the study is to compare the efficacy of levosimendan with that of dobutamine in patients with unstable hemodynamics (shock).

ELIGIBILITY:
Inclusion Criteria:

* Reduced left ventricular systolic function
* Hypotension
* Anuria or oligouria

Exclusion Criteria:

* Less than 18 years old
* Pregnant
* Uncorrected valvular stenosis
* Hypertrophic obstructive cardiomyopathy (HOCM)
* Third degree AV block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-10; Study Completion 2006-04

PRIMARY OUTCOMES:
Resolution of shock state

SECONDARY OUTCOMES:
Change in cardiac functions

CONTACTS AND LOCATIONS:
Locations (1):
- Intensive Care Unit, Nepean Hospital, Penrith, New South Wales, Australia